CLINICAL TRIAL: NCT00427219
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of Ozarelix, in Patients With Lower Urinary Tract Symptoms(LUTS) Due to Benign Prostatic Hypertrophy (BPH)
Brief Title: The Safety and Efficacy of Ozarelix to Treat Men With Lower Urinary Tract Symptoms Due to Enlargement of the Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPI-153-06-1
Record Dates: First submitted 2007-01-24; First posted 2007-01-26 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Benign Prostatic Hypertrophy
Keywords: Benign Prostatic Hyperplasia; Prostatic Adenoma, Benign; Prostatic Hypertrophy, Benign; Enlarged Prostate; Prostatism; Adenoma, Prostatic
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatism | interventions — ozarelix

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ozarelix (Experimental): All participants completing the placebo run in period were randomized to enter the treatment phase of the study and received ozarelix on Day 0 and Day 14.
  Interventions: Drug: Ozarelix
- Placebo (Placebo Comparator): All participants completing the placebo run in period were randomized to enter the treatment phase of the study and received placebo Day 0 and Day 14.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ozarelix — Ozarelix 15 mg will be administered IM on Day 0 and Day 14.
  Arms: Ozarelix
Drug: Placebo — Placebo will be administered IM on Day 0 and Day 14.
  Arms: Placebo

SUMMARY:
This study is to compare the efficacy and safety of ozarelix 15 mg given intramuscular (IM) 2 weeks apart on the improvement of symptoms and the duration of improvement for up to 6 months in men with Benign Prostatic Hypertrophy (BPH) who are over 50 years of age.

DETAILED DESCRIPTION:
This study is to compare the improvement in symptom scores, peak flow rate and quality of life in men suffering from lower urinary tract symptoms (LUTS) secondary to Benign Prostatic Hypertrophy (BPH) following treatment with ozarelix. Ozarelix is compared to placebo and injections given 14 days apart. Patients are followed for 6 months and both safety and efficacy assessed at monthly visits. Additionally, the impact of treatment on erectile function, if any, as well as Prostate-Specific Antigen (PSA) and Testosterone levels will be monitored.

The screening period of 7 days. The duration of the study is 40 weeks, including a 28-day placebo run-in phase (eligible participants entered a placebo run-in phase in which placebo is administered twice over a 2 week period [Day -28 and Day -14] and participants are assessed to establish baseline values approximately 14 days following the second placebo injection), study drug is administered on Days 0 and 14 followed by 34 weeks of observation after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

- All of the following questions must be answered "Yes" at Visit 1 in order for the participant to participate in the study.

* Is the participant at least 50 years old?
* Does the participant have clinical signs and symptoms consistent with BPH?
* Does the participant have an IPSS 13 at screening (prior to placebo run in)?
* Does the participant have a peak urinary flow rate (Qmax) of 4-15 milliliter/second (mL/sec) established on a voided volume of at least 125 mL?
* Is the participant willing to agree not to use any other approved or experimental pharmacologic BPH treatments including alpha blockers, 5-alpha reductase inhibitors, anti-cholinergic preparations or herbal preparations at any time during the study?

Exclusion Criteria: All of the following questions must be answered "No" at Visit 1 in order for the participant to participate in the study.

* Does the participant have a history of prostate cancer or a serum PSA >10 nanograms per milliliter (ng/mL)?
* Has the participant had prior prostate or bladder surgery, pelvic surgery (excluding hernia repair), pelvic radiation or lower urinary tract malignancy?
* Does the participant have a prevoid total bladder volume assessed by ultrasound > 550 mL?
* Does the participant have a residual urine volume > 350 mL by ultrasound?

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-01-23 (Actual); Primary Completion 2008-02-27 (Actual); Study Completion 2008-02-27 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in International Prostate Symptom Score (IPSS) | 12 weeks
  IPSS is a validated self-administered index for grading benign prostatic hyperplasia (BPH)-related signs and symptoms. It consists of a set of seven questions. A total score of 1-7 indicates mild disease, 8-19 moderate disease and 20-35 severe disease.

SECONDARY OUTCOMES:
International Prostate Symptom Score - Quality of Life (IPSS-QOL) | 36 weeks
  IPSS QOL is a disease-specific quality of life question, referred to as IPSS Question 8. Participants with an IPSS QOL of <3 at screening will be excluded from this study. The rating is as follows: 0=delighted, 1=pleased, 2=mostly satisfied, 3=mixed, 4=mostly dissatisfied, 5=unhappy, 6=terrible.
BPH Impact Index (BPHII) | 36 weeks
  BPH Impact Index (BII) is used to assess the impact of BPH on various aspects of health. This 4 question self administered index uses a scoring range from 0 (best) to 13 (worst).
Lower Urinary Tract Symptoms (LUTS) Global Assessment Question (LUTS-GAQ) | 36 weeks
  The self administered LUTS GAQ is a "yes" or "no" response to a question asking whether overall improvement in LUTS will be observed during the treatment period.
International Index of Erectile Function-15 (IIEF-15) | 36 weeks
  International Index of Erectile Function Erectile Function Domain (IIEF-EF) will be used to assess the effect of ozarelix on erectile function in sexually active men. IIEF-EF is defined as the sum of the scores for Questions 1-5 and 15 of the IIEF questionnaire. This recall instrument is self-administered by the participant. Individual questions are graded from 1 to 5 with a maximum total score of 30. Lower IIEF-EF scores represent diminished erectile function. Men with a score of ≥ 26 are interpreted as having normal erectile function.
Maximum Urinary Flow Rate (Qmax) | 36 weeks
  Qmax was measured by free flow uroflowmetry. Qmax is defined as the peak urine flow rate (measured in milliliter (mL)/second using a standard calibrated flowmeter). For a Qmax to be considered valid, the voided volume had to be at least 125 mL. The uroflowmeter is to be calibrated weekly.
Number of Participants With Adverse Events | 36 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Donald Gleason, MD, Tucson, Arizona
  - Jay Young, MD, Laguna Hills, California
  - Alexander Gershman, MD, Los Angeles, California
  - Stephen Auerbach, MD, Newport Beach, California
  - Eugene Dula, MD, Tarzana, California
  - Joel Kaufman, MD, Aurora, Colorado
  - Ira Klimberg, MD, Ocala, Florida
  - Joseph Williams, MD, Meridian, Idaho
  - Christopher Steidle, MD, Fort Wayne, Indiana
  - Steven Bigg, MD, St Louis, Missouri
  - Jed Kaminetsky, MD, New York, New York
  - William Fitch, MD, San Antonio, Texas
  - Gregg Eure, MD, Virginia Beach, Virginia